CLINICAL TRIAL: NCT05886114
Title: A Multi-domain Lifestyle Intervention Among Aged Community-residents in Zhejiang, China
Acronym: HERITAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xin Xu, Prof., Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 31005808A111272274170
Record Dates: First submitted 2023-05-08; First posted 2023-06-02 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Impairment; Alzheimer Disease; Vascular Cognitive Impairment; Dement; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorder; Cognition Disorder
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurocognitive Disorders; Mental Disorders; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Multi-domain Intervention (Experimental): Multi-domain structured intervention will be tailored by Chinese traditional and social norms and then conducted among the intervention group. That includes: Nutritional and dietary instruction, Cognitive training, Physical exercises, and Vascular risks monitoring and control.
  Interventions: Behavioral: Structured Multi-domain Intervention
- Self-Guided Intervention (Experimental): Every 6-12 months, control group will receive a regular health education campaign to encourage a healthy lifestyle and a regular health monitoring and examination of blood pressure, weight, fasting blood glucose and liposome group
  Interventions: Behavioral: Self-Guided Intervention

INTERVENTIONS:
Behavioral: Structured Multi-domain Intervention — Structured Multi-domain Intervention (SMI) involves providing participants with intensive structure and support by a team of trainers to increase physical exercise, adhere to a healthy diet, cognitive training, increase intellectual/social stimulation, and better manage vascular risk factors.
  Other Names: SMI
  Arms: Structured Multi-domain Intervention
Behavioral: Self-Guided Intervention — In the Self-Guided Intervention (SGI), education about the importance of a healthy lifestyle as a preventive strategy and support to encourage change will be provided.
  Other Names: SGI
  Arms: Self-Guided Intervention

SUMMARY:
A study conducted in Finland discovered that a multidomain intervention, consisting of physical activity, nutritional guidance, cognitive training, social activities, and management of vascular risk factors, effectively decelerated cognitive decline in healthy older adults who were at an increased risk of cognitive decline. The HERITAGE study is a 2-year clustered randomized controlled trial (clustered-RCT) that explores the efficacy of a multidomain intervention among 1200 elderly residents with a higher risk of cognitive decline and dementia in Zhejiang Province, China

DETAILED DESCRIPTION:
The effectiveness of a multidomain lifestyle intervention on the prevention of cognitive decline and dementia have not been studied in Asian elderly at high risk of dementia conversion. Dementia is caused by both nonmodifiable genetic variables, and modifiable lifestyle risk factors. While neuroimaging biomarkers have been well documented in the neurophysiology of ageing and age-associated cognitive decline, their role as surrogate endpoints and intermediate variables between multi-domain lifestyle intervention and cognitive benefits has not been studied. The current study aims to understand brain functional and structural changes that may result from a multi-domain lifestyle intervention and whether the changes correlate with improvement in cognitive function. At risk elderly aged 60-80 years will be randomly allocated to either the control arm (self-guided management) or the intervention (multi-domain lifestyle) arm, which consists of nutritional guidance, physical exercise, cognitive training and the monitoring and management of vascular and metabolic risk factors. We hypothesize that the multi-domain lifestyle intervention will promote favorable changes in cognitive function. Moreover, such intervention will slow down the progression of cerebrovascular disease and neurodegeneration in participants in the intervention arm. Findings from the present study will shed light on the biological mechanisms of age-related cognitive decline and neurodegenerative disease. Insight obtained from the study could be translated into new targets of nonpharmacological interventions which aim at the potential causal molecular pathways implicated in ageing and age-related cognitive decline. Adaption and implementation of our findings into clinical and public health practice will further promote healthy and confident ageing among Chinese elderly, to eventually expand their health span.

ELIGIBILITY:
Inclusion Criteria:

* At risk of cognitive decline: cognitive performance at the mean level or slightly lower than expected for age with no dementia (AD8>=3 and/or 5-min MoCA >, < 11)
* Free of physical disabilities that preclude participation in the study
* Willing to complete all study-related activities for 24 months
* Willing to be randomized to either lifestyle intervention group

Exclusion Criteria:

* Diagnosed dementia patients
* Diagnosed major depression or other neuropsychological diseases
* Malignant diseases
* Symptomatic cardiovascular disease
* Revascularization within one year
* Severe loss of vision, hearing or communicative ability

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2023-05-28 (Estimated); Primary Completion 2025-04-28 (Estimated); Study Completion 2027-04-28 (Estimated)

PRIMARY OUTCOMES:
Global Cognition | Up to 2 years
  Globe cognitive performance (composite z-score) measured by comprehensive Neuropsychological Test Battery (NTB)
Domain-specific Cognition | Up to 2 years
  NTB domain-specific cognitive performance (composite z-score) for memory, executive function, attention, language, visuomotor speed and visuoconstruction.

SECONDARY OUTCOMES:
Neuroimaging: MRA | Up to 2 years
  Changes in brain blood flow assessed by magnetic resonance angiography(MRA)
Neuroimaging: MRI | Up to 2 years
  Changes in brain structural integrity (gray matter volume loss, white matter microstructure degradation and increase of cerebrovascular markers) assessed by T1-weighted Magnetization Prepared Rapid Gradient Recalled Echo, Fluid Attenuated Inversion Recovery (FLAIR), T2-weighted, and Susceptibility Weighted Imaging sequences
Neuroimaging: fMRI | Up to 2 years
  Changes in brain functional networks assessed by fMRI
Number of participants with Laboratory Values /Blood markers | Up to 2 years
  Blood samples will be collected from all patients in tubes with ethylenediaminetetraacetic acid 0.1%. Changes in Novel and accessible blood markers to monitor AD- and CeVD- associated pathologies. Plasma concentrations of cardiac markers (High-sensitive cardiac troponin T (hs Troponin T), N-terminal pro b-type natriuretic peptide (NT-proBNP) and Growth/differentiation factor 15 (GDF 15)), and peripheral biomarkers of Aβ, tau and synaptic pathology, oxidative stress, endothelial/cardiovascular injury and degenerative protein modifications (DPMs) damaged proteins will be measured by laboratory testings.
Incident dementia | Up to 2 years
  Incidence of dementia. Dementia diagnoses will be made by CDR and DSM-IV criteria.
Clinical Dementia Rating-Sum of Boxes (CDR-SB) | Up to 2 years
  The Clinical Dementia Rating-Sum of Boxes (CDR-SB) is scored from 0 to 18. Higher scores reflect worse performance.
Alzheimer's Disease Cooperative Study Activities of Daily Living Mild Cognitive Impairment-Activities of Daily Living Inventory (ADCS MCI-ADL) | Up to 2 years
  The Alzheimer's Disease Cooperative Study Activities of Daily Living-Mild Cognitive Impairment-Activities of Daily Living Inventory (ADCS MCI-ADL) is scored from 0 to 53. Higher scores reflect better performance.
Cardiovascular morbidity | Up to 2 years
  Physician-diagnosed cardiometabolic health disorders will be identified based on ICD-9 or ICD-10 codes (in any position). Any incident cardiometabolic morbidity, for example, ardiac dysrhythmias, heart failure, peripheral and visceral atherosclerosis, non-alcoholic fatty liver disease, chronic kidney disease, type 2 diabetes, hypercholesterolemia, and hypertension, will be recorded.
Physical Performance: Grip strength | Up to 2 years
  Grip strength will be assessed by a hydraulic hand dynamometer and expressed in absolute units(kilograms) andrelative units(kilograms divided by bodyweight).
Physical Performance: Gaid speed | Up to 2 years
  Walking pace will be assessed by the speed (m/second) of completing a 1.5 meters walk.
Physical Performance: Balance | Up to 2 years
  Balance will be measured by standing on one foot and expressed in absolute units(seconds).
Physical Performance: Endurance | Up to 2 years
  Endurance will be assessed by the 2MW. Participants will be asked to "walk as fast as you can without running" for 2 minutes around a 50-foot course. A greater distance(m) indicates better endurance.
Physical Performance: Lower limb strength | Up to 2 years
  Lower limb strength will be assessed by 30 second sit to stand test and expressed by completion times.
Quality of Life Questionnaire (15D) | Up to 2 years
  The Quality of Life Questionnaire (15D) has a single index (15D score) on a 0-1 scale, which represents overall HRQoL (0 = being dead, 0.0162 = being unconscious or comatose, 1 = no problems on any dimension = 'full' HRQOL). This is calculated from the health state descriptive system by using a set of population-based preference or utility weights.
The Geriatric Depression Scale (GDS) | Up tp 2 years
  The Geriatric Depression Scale (GDS) is scored from 0 to 15. Scores of 0-4 are considered normal, 5-8 indicate mild depression; 9-11 indicate moderate depression; and 12-15 indicate severe depression.
Pittsburgh Sleep Quality Index (PSQI) | Up to 2 years
  The Pittsburgh Sleep Quality Index (PSQI) is scored from 0 to 21. Higher scores indicate worse sleep quality.
Leisure-Time Activities Questionnaire | Up to 2 years
  The Leisure-Time Activities Questionnaire measures the frequency of engagement in the following activities: Health activities, Social activities, Productive activities, Fitness activities, Recreational activities, Any cognitively-stimulating activities. Scores are measured on a 3-point scale. Higher scores represent higher frequency of engagement in leisure-time activities.
Resource Use Inventory (RUI) | Up to 2 years
  The Resource Use Inventory (RUI) measures 4 domains: direct medical care, direct nonmedical care, informal care, and subjects' time use. The RUI is filled in based on the frequency and amount of resources used. If none were used, '00' is entered.
Hight | Up to 2 years
  Height will be measured in metres
Weight | Up to 2 years
  Weight will be measured in kilograms.
Hip circumference | Up to 2 years
  Hip circumference will be measured in centimetres.
Waist circumference | Up to 2 years
  Waist circumference will be measured in centimetres.
Changes in Blood Pressure | Up to 2 years
  Vascular and metabolic risk factors measured by changes in blood pressure in mmHg. Incident events using serious adverse event reports will also be assessed.
Changes in lipid Profile | Up to 2 years
  Blood samples will be collected from all patients in tubes with ethylenediaminetetraacetic acid 0.1%. Lipid Profile will be expressed by total cholesterol, LDL-cholesterol, HDL-cholesterol or triglycerides in mmol/L.
Changes in Glucose Regulation | Up to 2 years
  Vascular and metabolic risk factors measured by changes in glucose regulation in mmol/L.
Retinal Imaging Markers | Up to 2 years
  Retinal fundus photographs will be taken of each eye with a nonmydriatic digital camera after dilation of pupils with 1% tropicamide eye drops. A semi-automated computer-assisted program will be used to assess retinal vascular fractal dimensions (among other parameters such as vessel caliber and vessel tortuosity) from optic disc-centered images of a randomly selected eye per participant.
Falls | Up to 2 years
  Prospective rate of falls, causes and consequences via monthly calendar will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health and The Second Affiliated Hospital of School of Medicine, Zhejiang University, Hangzhou, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Interested collaborators may put in a request.

REFERENCES:
- [Background] Xu X, Chew KA, Wong ZX, Phua AKS, Chong EJY, Teo CKL, Sathe N, Chooi YC, Chia WPF, Henry CJ, Chew E, Wang M, Maier AB, Kandiah N, Chen CL. The SINgapore GERiatric Intervention Study to Reduce Cognitive Decline and Physical Frailty (SINGER): Study Design and Protocol. J Prev Alzheimers Dis. 2022;9(1):40-48. doi: 10.14283/jpad.2022.5. PMID 35098972
- [Result] Zhao X, Hu R, Wen H, Xu G, Pang T, He X, Zhang Y, Zhang J, Chen C, Wu X, Xu X. A voice recognition-based digital cognitive screener for dementia detection in the community: Development and validation study. Front Psychiatry. 2022 Jul 22;13:899729. doi: 10.3389/fpsyt.2022.899729. eCollection 2022. PMID 35935417